CLINICAL TRIAL: NCT00004457
Title: Determinants of Disease Severity in Amyotrophic Lateral Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Massachusetts General Hospital (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/13650; MGH-97-7231; MGH-1K08NS01896
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; motor neuron disease; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
OBJECTIVES:

I. Determine specific clinical features, molecular abnormalities, and laboratory-based biological markers of free radical stress that are associated with amyotrophic lateral sclerosis and influence disease severity.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a screening and diagnostic study. Blood and urine samples are collected from patients every 2 months for 1 year. All samples are evaluated for measures of free radical damage and levels of the body's own antioxidant activity.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Clinically diagnosed probable or definite, sporadic or familial amyotrophic lateral sclerosis

--Patient Characteristics-- Pulmonary: No artificial ventilation required Other: No other neurodegenerative diseases No concurrent or history of unstable medical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: Merit E. Cudkowicz, Study Chair — Massachusetts General Hospital